CLINICAL TRIAL: NCT06452342
Title: TRanEXamic Acid to Decrease Heavy Menstrual Bleeding in Individuals Anticoagulated for Venous Thromboembolism Pilot Study
Acronym: T-REX HMB
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network)
Responsible Party: Principal Investigator, Jameel Abdulrehman, Staff Hematologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-5178.0
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Venous Thromboembolism; Venous Thromboses; Heavy Menstrual Bleeding; Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Menorrhagia; Hemostatic Disorders | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (Experimental): Tranexamic acid (Cyclokapron®) 1.5 grams, orally, three times a day during menstrual cycle for the 3 month study period.
  Interventions: Drug: Tranexamic acid
- No tranexamic acid (Other): Routine clinical care without Tranexamic acid
  Interventions: Other: No Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid 1.5 grams, orally, three times a day during menstrual cycle for the 3 month study period
  Other Names: Cyclokapron
  Arms: Tranexamic acid
Other: No Tranexamic acid — Routine clinical care without Tranexamic acid
  Arms: No tranexamic acid

SUMMARY:
T-REX HMB is a pilot randomized controlled trial (RCT) designed to assess the feasibility of a full trial comparing tranexamic acid (TXA) to placebo in decreasing HMB in premenopausal individuals anticoagulated for VTE. Strong data supports TXA as an effective and safe agent at decreasing HMB in the general population, but its use in those with VTE has been limited by a lack of data for its efficacy in anticoagulated individuals and theoretical concerns of its prothrombotic effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult pre-menopausal individuals with regular menstrual cycles (defined as menstrual bleeding every 24 to 38 days)
2. Diagnosed with acute VTE on objective imaging;
3. Within two weeks of starting treatment with therapeutic dose anticoagulation;
4. Planned treatment of at least 3 months of therapeutic dose anticoagulation.
5. Written informed consent in accordance with federal, local and institutional guidelines.

Exclusion Criteria:

1. Hypersensitivity or allergy to TXA
2. Active major bleeding other than menstrual bleeding
3. Use of hormonal contraceptives
4. Known history of thrombosis and antiphospholipid syndrome (including those patients that are triple positive for lupus anticoagulant, anticardiolipin antibodies, and anti-beta 2-glycoprotein I antibodies.
5. Known renal insufficiency
6. Pregnant or breastfeeding
7. Use of other thrombotic agents
8. Under 18 years of age
9. Patient is unable to provide informed consent (lacking capacity, language etc)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment to study | 3 months
  Number of participants successfully recruited to the study and randomized to a treatment arm

SECONDARY OUTCOMES:
Participant adherence to the study drug | 3 months
  Defined as the proportion of menstrual days in which TXA was taken
Participant compliance with study procedures | 3 months
  Defined as >75% study drug adherence and no missed follow up visits
Loss to follow-up or drop-out | 3 months

OTHER OUTCOMES:
Menstrual blood loss per menstrual cycle | 3 months
  Measured by the pictorial blood loss assessment chart (PBAC).
  The PBAC has a minimum value of 0 and no maximum value, with a higher score indicating a worse outcome.
Menstrual blood loss in days | 3 months
  Menstrual blood loss in days, over total study follow up time;
Menstrual blood loss in days with PBAC > 5 | 3 months
  Menstrual blood loss in days with PBAC > 5, over total study follow up time
Major bleeding events | 3 months
  As defined by the International Society on Thrombosis and Haemostasis (ISTH)
Clinically relevant non-major bleeding | 3 months
  As defined by the International Society on Thrombosis and Haemostasis (ISTH)
Ferritin | 3 months
  Ferritin blood work
Hemoglobin | 3 months
  Hemoglobin blood work
Recurrent venous thromboembolism | 3 months
  Objectively confirmed on appropriate diagnostic imaging
Symptoms of post thrombotic syndrome | 3 months
  Symptoms of post thrombotic syndrome at 3 months using the Venous Insufficiency Epidemiological and Economic Study - Quality of Life (VEINES-QOL) survey in those with previous DVT.
  The VEINES-QOL survey has a minimum value of 0 and a maximum value of 118, with a higher score indicating a better outcome.
QOL after PE | 3 months
  QOL (quality of life) after PE at 3 months using the PEmb-QOL (Pulmonary Embolism - Quality of Life) survey in those with previous PE.
  The PEmb-QOL survey has a minimum value of 0 and a maximum value of 100, with a higher score indicating a worse outcome.
General health related QOL | 3 months
  General health related QOL using the Short Form Health Survey (SF-36).
  The SF-36 has a minimum value of 0 and a maximum value of 100 per health domain, with a higher score indicating a better outcome.

IPD SHARING:
Plan to Share IPD: No